CLINICAL TRIAL: NCT04750044
Title: Timing of Oral Refeeding in Post-ERCP Pancreatitis
Brief Title: Refeeding in Post-ERCP Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2020-1237
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Post-ERCP Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early refeeding group (Experimental): In the early refeeding group, oral diet is started 24 hours after PEP is confirmed.
  Interventions: Other: early refeeding
- delayed refeeding group (Active Comparator): In the delayed refeeding group, oral diet is started after confirmation of restoring of normal bowel sound, pain decreasing below VAS 2.
  Interventions: Other: delayed refeeding

INTERVENTIONS:
Other: early refeeding — In the early refeeding group, oral diet is started 24 hours after PEP is confirmed. The oral diet starts with SOW (Sips of water) and builds up sequentially in the order of clear liquid diet-soft diet, considering patient tolerability.
  Arms: early refeeding group
Other: delayed refeeding — In the delayed refeeding group, oral diet is started after confirmation of restoring of normal bowel sound, pain decreasing below VAS 2. The oral diet starts with SOW (Sips of water) and builds up sequentially in the order of clear liquid diet-soft diet, considering patient tolerability.
  Arms: delayed refeeding group

SUMMARY:
Endoscopic retrograde cholangio-pancreatography (ERCP) is the most commonly used technique for diagnosis and treatment in the treatment of bile duct diseases including bile duct cholelithiasis and malignant/benign biliary obstruction. In particular, ERCP is an essential procedure for the removal of bile duct gallstones and bile drainage in malignant/benign biliary obstruction patients.

Among ERCP-related complications, especially "post-ERCP pancreatitis (PEP)", which occurs due to the anatomical structure of the pancreatic biliary system, statistically occurs in about 5-10% of patients who first received ERCP. It is known, and treatment for PEP is the same as treatment for general acute pancreatitis but is known to have a relatively worse prognosis.

The basis of treatment for acute pancreatitis is a conservative treatment based on fasting and fluid treatment, and starting oral diet after abdominal pain and pancreatic enzyme levels (amylase/lipase) normalized. However, a recent study reported that early oral diet could improve the patient's prognosis. According to a systematic review of 11 randomized trial papers by Valerie et al., it was reported that the early diet had the effect of reducing hospital stay without increasing adverse events when comparing the prognosis of the early refeeding group and delayed refeeding group. This result is theoretically considered to be because the oral diet has the advantage of increasing intestinal permeability, gut motility and reducing the likelihood of pancreatic necrosis/ infection compared to the parenteral diet.

As above, PEP has the same treatment method as general acute pancreatitis but is known to have a relatively worse prognosis. However, the effect of an early diet recently attempted in acute pancreatitis has not been reported in patients with PEP. Therefore, we investigate the effects of early and delayed diets on the prognosis of patients with PEP through a prospective multicenter study.

DETAILED DESCRIPTION:
1. Selection of research subjects A total of 80 patients, who have occurred pancreatitis after ERCP, will be enrolled at Yonsei University Sinchon Severance Hospital, Seoul National University Hospital, Dongguk University Ilsan Hospital, Gachon University Gil Hospital, Gyeongsang National University Changwon Hospital, Kyungpook National University Hospital, Seoul St. Mary's Hospital, Korea University Ansan Hospital, Pusan National University Hospital. The purpose and contents of this clinical trial are informed in detail to the subject and consent is obtained.
2. Evaluation of eligibility Eligibility is determined based on the basic patient data including physical examination, vital signs, body measurements, medical history, concomitant drugs, laboratory tests, and other basic examinations made at the first visit.
3. Grouping and randomization After ERCP was performed, the study subjects who were judged to have PEP according to enroll criteria were divided into early and delayed refeeding groups using a random number table and assigned 1:1 to proceed with the study.
4. Timing of refeeding In the early refeeding group, oral diet is started 24 hours after PEP is confirmed.

   In the delayed refeeding group, oral diet is started after confirmation of restoring of normal bowel sound, pain decreasing below VAS 2. The oral diet starts with SOW (Sips of water) and builds up sequentially in the order of clear liquid diet-soft diet, considering patient tolerability.
5. Interruption of refeeding In both early and delayed refeeding groups, the oral diet is stopped when the pain scale the patient complains after starting oral diet increases to VAS 5 points or more, or the patient refuses to eat due to abdominal pain or other reasons. The diet is restarted after the amylase/lipase level decreases below the upper normal limit, the patient's pain has disappeared, and the bowel movement is restored.
6. Dropout criteria

   1. In the case of delayed diet group when symptoms persist for more than 96 hours and cannot start a diet
   2. When fasting is necessary for other reason, such as an imaging test or endoscopy
   3. When it is determined that a parenteral diet is necessary for reasons such as difficulty swallowing
   4. When the researcher judged that the clinical trial cannot be continued
7. Discharge criteria and hospitalization period for PEP If the patient is tolerable for more than 24 hours after the soft diet (abdominal pain improvement, lab amylase/lipase level decreases to less than 2 times the upper normal limit, it is judged that PEP has improved and the discharge criteria have been satisfied. From the point of diagnosis of PEP to the point of time when the discharge criteria are satisfied is defined as the "hospitalization period for PEP".

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 to 80
2. As patients who developed pancreatitis after receiving ERCP, the following must be satisfied at the same time.

   1. increased serum amylase or lipase 3 times higher than the normal range, at 4 hours after ERCP or the morning of the following day,
   2. New or worsening abdominal pain compatible with pancreatitis, arising 4 hours after ERCP or the next morning

Exclusion Criteria:

1. If the intended procedure is not completed
2. If complications such as abdominal perforation or bleeding have occurred or are suspected
3. If it is judged as severe acute pancreatitis with multi-organ failure la.
4. When PEP has occurred, but additional imaging tests and endoscopy for diagnosis of the underlying disease or treatment of complications of the patient are required, and fasting is necessary regardless of this study
5. Patients with a history of chronic pancreatitis
6. Pregnant women, lactating women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
hospitalization period for PEP | up to 1 month
  If the patient is tolerable for more than 24 hours after the soft diet (abdominal pain improvement, lab amylase/lipase level decreases to less than 2 times the upper normal limit, it is judged that PEP has improved and the discharge criteria have been satisfied. From the point of diagnosis of PEP to the point of time when the discharge criteria are satisfied is defined as the "hospitalization period for PEP".

SECONDARY OUTCOMES:
Incidence of acute severe pancreatitis | up to 1 month
  comparing rate of incidence of severe acute pancreatitis
readmission rate (<30 days) | up to 1 month
  comparing readmission rate of each group until 30 days after discharge
mortality rate | up to 1 month
  comparing mortality rat of each group during hospitalization
complication rate | up to 1 month
  comparing complication rate including nausea/vomiting, recurrent abdominal pain, necrotizing pancreatitis of each group during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hyun Jo, Principal Investigator — Severance Hospital
Locations (9):
- South Korea (9):
  - Korea University Ansan Hospital, Ansan-si
  - Pusan National University Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Kyungpook National University School of Medicine, Daegu
  - Gachon University College of Medicine, Incheon
  - Yonsei University College of Medicine, Seoul
  - Seoul Metropolitan Government Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jo JH, Lee JM, Jang DK, Choe JW, Han SY, Choi YH, Kim EJ, Kim HY, Jung MK, Lee SH. Early Oral Refeeding in Patients with Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis: A Randomized Controlled Trial. Gut Liver. 2025 Nov 15;19(6):900-908. doi: 10.5009/gnl250110. Epub 2025 Aug 25. PMID 40852738